CLINICAL TRIAL: NCT02254213
Title: Intra-individual Stability in EEG Parameters
Brief Title: Intra-individual Stability in Electroencephalography (EEG) Parameters
Status: Completed | Type: Observational
Sponsor: Mentis Cura (Industry)
Collaborators: The Icelandic Center for Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: MC-CT-003
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Stability of EEG Features in Humans
Keywords: Intra-individual stability, EEG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: EEG recording — A short EEG recording is performed 10 times over the span of three months.

SUMMARY:
The main objective is to evaluate the stability of EEG features on an individual level.

ELIGIBILITY:
Inclusion Criteria:

* Age must be in the range 50 - 90 years

Exclusion Criteria:

* Outside required age range

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 15 individuals in the age range of 50 - 90 years.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2005-06; Primary Completion 2005-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Quantitative EEG (qEEG) features | Three months
  qEEG features are extracted from 10 separate EEG recordings from each individual in the cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Kristinn Johnsen, PhD, Principal Investigator — Mentis Cura

REFERENCES:
- [Result] Gudmundsson S, Runarsson TP, Sigurdsson S, Eiriksdottir G, Johnsen K. Reliability of quantitative EEG features. Clin Neurophysiol. 2007 Oct;118(10):2162-71. doi: 10.1016/j.clinph.2007.06.018. Epub 2007 Aug 31. PMID 17765604